CLINICAL TRIAL: NCT01332721
Title: An Open Label Phase 1B Dose-Escalation Study of TRC105 Combined With Standard-Dose Bevacizumab for Advanced Solid Tumors
Brief Title: Study of TRC105 Combined With Standard-Dose Bevacizumab for Advanced Solid Tumors for Which Bevacizumab is Indicated
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tracon Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 105ST102
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Results first posted 2014-03-28 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-11

CONDITIONS: Adult Solid Tumor
Keywords: TRC105; CD105; Endoglin; Solid Tumors; Avastin; Bevacizumab
MeSH Terms: interventions — carotuximab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TRC105 and Bevacizumab (Experimental): Escalating doses of i.v. TRC105 will be administered weekly beginning with 3 mg/kg in combination with 15 mg/kg bevacizumab given every 3 weeks. Patients will receive TRC105 treatment on Days 1, 8, and 15 and bevacizumab treatment on Day 1 of each 21-day cycle.
  Interventions: Drug: TRC105 and Bevacizumab

INTERVENTIONS:
Drug: TRC105 and Bevacizumab — Escalating doses of i.v. TRC105 will be administered weekly beginning with 3 mg/kg in combination with 15 mg/kg bevacizumab given every 3 weeks. Patients will receive TRC105 treatment on Days 1, 8, and 15 and bevacizumab treatment on Day 1 of each 21-day cycle.
  Other Names: Chimeric Antibody (TRC105) to CD105; Avastin

SUMMARY:
The purpose of the study is to evaluate safety and tolerability and determine a recommended Phase 2 dose for TRC105 when added to standard dose bevacizumab in patients with advanced solid tumors for which bevacizumab is indicated.

DETAILED DESCRIPTION:
Bevacizumab is a monoclonal antibody to vascular endothelial growth factor (VEGF) that inhibits angiogenesis and extends survival in patients with a wide variety of solid tumor types. TRC105, a monoclonal antibody to CD105, is a novel angiogenesis inhibitor that complements bevacizumab in preclinical models. Together, these antibodies may result in more effective angiogenesis inhibition and improved clinical efficacy over that seen with bevacizumab alone. The purpose of the study is to evaluate safety and tolerability and determine a recommended Phase 2 dose for TRC105 when added to standard dose bevacizumab in patients with advanced solid tumors for which bevacizumab is indicated.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven advanced or metastatic solid cancer
2. Measurable disease, evaluable disease or elevation of a relevant soluble tumor marker (e.g., CEA, PSA, CA125)
3. Age of 18 years or older
4. ECOG performance status of 0 or 1
5. Resolution of all acute AEs resulting from prior cancer therapies to NCI CTCAE Grade ≤ 1 or baseline (except alopecia)
6. Adequate organ function
7. Willing and able to consent for self to participate in study

Exclusion Criteria:

1. Prior treatment with TRC105
2. Serious dose-limiting toxicity related to prior bevacizumab
3. Current treatment on another therapeutic clinical trial
4. Receipt of an investigational agent within 28 days of starting study treatment
5. Prior surgery (including open biopsy) within 28 days of starting the study treatment
6. Prior radiation therapy or systemic therapy within 21 days of starting the study treatment
7. Minor surgical procedures such as fine needle aspirations, Mediport placement or core biopsies within 7 days of study treatment
8. Uncontrolled chronic hypertension defined as systolic > 140 or diastolic > 90 despite optimal therapy (initiation or adjustment of BP medication prior to study entry allowed provided that the average of 3 BP readings at a visit prior to enrollment is < 140/90 mm Hg)
9. Symptomatic pericardial or pleural effusions
10. Uncontrolled peritoneal effusions requiring paracentesis more frequently than every 2 weeks
11. History of brain involvement with cancer, spinal cord compression, or carcinomatous meningitis, or new evidence of brain or leptomeningeal disease (except in the expansion cohort at the MTD where brain metastases or primary brain tumors are eligible)
12. Angina, MI, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, arterial embolism, pulmonary embolism, DVT, PTCA or CABG within the past 6 months
13. Active bleeding or pathologic condition that carries a high risk of bleeding
14. Thrombolytic or anticoagulant use (except to maintain i.v. catheters) within 10 days prior to first day of study therapy
15. Cardiac dysrhythmias of NCI CTCAE Grade ≥ 2 within the last 28 days
16. Known active viral or nonviral hepatitis
17. Centrally located non-small cell lung cancer (regardless of histologic sub-type), or non-small cell lung cancer of squamous histology.
18. History of hemorrhage or hemoptysis (>½ teaspoon bright red blood) within 6 months of starting study treatment
19. Open wounds or unhealed fractures within 28 days of starting study treatment
20. History of peptic ulcer disease or erosive gastritis within the past 6 months, unless treated for the condition and complete resolution has been documented by esophagogastroduodenoscopy (EGD) within 28 days of starting study treatment
21. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness
22. Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-04; Primary Completion 2012-09 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles P Theuer, MD, Study Director — Tracon Pharmaceuticals Inc.
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Pinnacle Oncology Hematology, Scottsdale, Arizona
  - UCLA Hematology and Oncology, Santa Monica, California
  - Indiana University Simon Cancer Center, Indianapolis, Indiana

RESULTS

PARTICIPANT FLOW:
Groups:
- TRC105 and Bevacizumab: Escalating doses of TRC105 were studied in combination with standard dose bevacizumab. In accordance with the original protocol, patients in cohorts 1 and 2 received TRC105 on day 1, day 8, and day 15 and bevacizumab on day 1 of each 3 week cycle. Cohort 3 and 4 patients received TRC105 on days 8, 15, and 22 and bevacizumab on days 1 and 15 of cycle 1 (4 week cycle), and cohort 4a and 5 patients received TRC105 on days 8, 11, 15, and 22 and bevacizumab on days 1 and 15 of cycle 1 (4 week cycle). Beyond cycle 1, patients in cohorts 3, 4, 4a, and 5 received TRC105 on days 1, 8, 15 and 22 and bevacizumab on days 1 and 15 of each 4 week cycle.
Period: Overall Study
Arm/Group | TRC105 and Bevacizumab
Started | 38
Completed | 38
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TRC105 and Bevacizumab
Number analyzed (Participants) | 38
Age, Continuous [Median (Full Range); unit: Years] | 63 [42 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 15
Prior VEGF inhibitor treatment [Number; unit: participants]
  Prior VEGF inhibitor treatment | 30
  No prior VEGF inhibitor treatment | 8

OUTCOME MEASURES:

1. Primary Outcome: Determine Maximum Tolerated Dose of TRC105 in Combination With Bevacizumab
Description: Three patients will be initially enrolled and treated at each dose level. If none of these 3 patients experiences a dose-limiting toxicity (DLT) during the 28-day evaluation period, dose escalation will proceed following review of safety data with appropriate site staff including the principal investigators at all sites. If 1 of 3 patients experiences DLT, the cohort will be expanded to 6 patients. The maximum tolerated dose (MTD) will have been exceeded if ≥ 33% of patients experience DLT in a given cohort. DLT will have occurred when a patient has 1 or more toxicity listed in the table below that is at least possibly related to the combination of bevacizumab and TRC105 during the first 28 days (cycle 1).
Time Frame: 1.5 years
Measure: Number; unit: mg/kg
Arm/Group | TRC105 and Bevacizumab
Number analyzed (Participants) | 38
mg/kg | 10

2. Secondary Outcome: TRC105 Pharmacokinetic Concentrations
Description: Plasma TRC105 concentrations will be measured at specified timepoints.
Time Frame: 1.5 years
Reporting Status: Not Posted

3. Secondary Outcome: Immune Response to TRC105
Description: HAMA and HACA titers will be measured at specified time-points.
Time Frame: 1.5 years
Measure: Number; unit: participants
Arm/Group | TRC105 and Bevacizumab
Number analyzed (Participants) | 26
participants
  HAMA POSITIVE | 3
  HAMA NEGATIVE | 23
  HACA POSITIVE | 4
  HACA NEGATIVE | 22

4. Secondary Outcome: Objective Response According to RECIST 1.1
Description: The best response according to RECIST 1.1 for each patient with measurable disease and who received at least one dose of study drug will be listed by cohort and tumor type
Time Frame: 1.5 years
Measure: Number; unit: participants
Arm/Group | TRC105 and Bevacizumab
Number analyzed (Participants) | 31
participants
  RECIST 1.1 defined response | 2
  Tumor burden decreases | 14

ADVERSE EVENTS:
Time Frame: The adverse event reporting period for this trial started when a given patient had the first dose of bevacizumab and/or TRC105 study drug and ended 28 days after the last dose of bevacizumab and/or TRC105 study drug was administered whichever was later. In addition, any known untoward event that occurred beyond the adverse event reporting period that the Investigator assessed as possibly related to TRC105 and/or bevacizumab was reported as an adverse event.
Arm/Group | TRC105 and Bevacizumab
Serious Adverse Events (participants affected / at risk) | 9/38
Other Adverse Events (participants affected / at risk) | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TRC105 and Bevacizumab (N=38)
Ileus (Gastrointestinal disorders) | 1 (1) — Not related to TRC105
Cellulitis of Left Foot (Infections and infestations) | 1 (1) — Not Related to TRC105
Recurrent pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Not Related to TRC105
Headache (Nervous system disorders) | 1 (1) — Suspected Adverse Reaction
disease progression (General disorders) | 1 (1) — Not Related to TRC105
Pneumonia (Infections and infestations) | 1 (1) — Not related to TRC105
MRSA Sepsis (Infections and infestations) | 1 (1) — Not Related to TRC105
Sepsis (Infections and infestations) | 1 (1) — not related to TRC105
Brain Absces (Infections and infestations) | 1 (1) — Suspected Adverse Reaction
Small Bowel Obstruction (Gastrointestinal disorders) | 1 (1) — Not Related to TRC105
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TRC105 and Bevacizumab (N=38)
Anaemia (Blood and lymphatic system disorders) | 11
Hypothyroidism (Endocrine disorders) | 2
Periorbital oedema (Eye disorders) | 2
Gingival pain (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 3
Oral pain (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Face oedema (General disorders) | 4
Fatigue (General disorders) | 10
Infusion related reaction (Injury, poisoning and procedural complications) | 11
Decreased appetite (Metabolism and nutrition disorders) | 4
Headache (Nervous system disorders) | 31
Migraine (Nervous system disorders) | 3
Sinus headache (Nervous system disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3
Epistaxis (Vascular disorders) | 25
Flushing (Vascular disorders) | 8
Gingival bleeding (Vascular disorders) | 12
Telangiectasia (Vascular disorders) | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less